CLINICAL TRIAL: NCT02876536
Title: Effect of Transcutaneous Electrical Nerve Stimulation on Cognitive Disorders in Multiple Sclerosis Patients
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation on Cognition in Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, assistant prof, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Isfahan MS society
Record Dates: First submitted 2016-08-14; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis; Cognitive Disorders
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNES with sending electrical impulses (Experimental): The MS patients will receive electrical impulses by TENS device for 30 minutes a day, for 5 days a week and in 6 weeks
  Interventions: Device: TENS
- TENS without sending electrical impulses (Sham Comparator): The MS patients will use the TENS device for 30 minutes a day, for 5 days a week and in 6 weeks without receiving any electrical impulses
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — The effect of TENS device will be compared in case and control groups.

SUMMARY:
The aim of this study is to evaluate whether the Transcutaneous Electrical Nerve Stimulation (TENS) is effective on improvement of cognitive disorders in Multiple sclerosis patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is one of the most common autoimmune diseases in the world. One of the complications of MS, is cognitive disorder.

In some studies on rats, stimulation of somatosensory neurons has improved the hippocampus activity by increasing the amount of acetylcholine. Hippocampus has a major role in cognition and behavior.

TENS is a non-invasive method in which the electrical pulses are sent to the body trough skin by electrodes. This device can stimulate the somatosensory neurons by electrical impulses. In several studies, the effect of TENS has been proved on short term memory and verbal fluency in patients with mild stages of Alzheimer disease. Also it has been effective on some aspects of cognition on old people suffering from forgetfulness.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed multiple sclerosis by McDonald criteria;
* score 25 or less in mini mental state examination (MMSE)

Exclusion Criteria:

* MMSE score greater than 25;
* the history of psychiatric problems;
* addiction to alcohol; head trauma; cerebrovascular disease; hydrocephalus; neoplasm; epilepsy; renal or respiratory diseases; impaired consciousness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
change in the level of cognition measured by Addenbrooke's cognitive examination | 6 weeks
  Addenbrooke's cognitive examination has 100 parts and measures different aspects of cognition including memory, concentration, language, verbal fluency and visuospatial skills. The patients will take the test before and after using the TENS device

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Shaygannezhad, professor, Study Director — Isfahan MS Society, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Alzahra Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided